CLINICAL TRIAL: NCT03393078
Title: Study of Brain Network Mechanism for Individualized Accurate Target Positioning rTMS Treatment on Obsessive Compulsive Disorder
Brief Title: Repetitive Transcranial Magnetic Stimulation (rTMS) Treatment for Obsessive Compulsive Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, Chunyan Zhu, A/Prof., Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AnhuiMU
Record Dates: First submitted 2017-12-28; First posted 2018-01-08 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Obsessive-Compulsive Disorder; Transcranial Magnetic Stimulation; Functional Magnetic Resonance Imaging; Event-Related Potentials
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Real Stimulation (Active Comparator): The repetition transcranial magnetic stimulation(rTMS) lasted 30 mins and delivered at 1 Hz with 1s duration, a total of 1800 pulses at 110% of the rest motor threshold (RMT) . MRI dataset should be acquired before the first rTMS session and after the last rTMS session.
  Interventions: Device: transcranial magnetic stimulation with real coil
- Sham Stimulation (Sham Comparator): The procedure of this protocol was performed by a placebo coil, lasted 30 mins and delivered at 1 Hz with 1s duration, a total of 1800 pulses at 110% of the rest motor threshold (RMT). No actual magnetic stimulation was applied on the head of the volunteers. MRI dataset should be acquired before the first rTMS session and after the last rTMS session.
  Interventions: Device: transcranial magnetic stimulation with sham coil

INTERVENTIONS:
Device: transcranial magnetic stimulation with real coil — TMS with real coil is a noninvasive technique to activate and modify the activity of the neurons
  Arms: Real Stimulation
Device: transcranial magnetic stimulation with sham coil — TMS with sham coil is a placebo
  Arms: Sham Stimulation

SUMMARY:
To investigate the treatment effect of repetitive transcranial magnetic stimulation on Obsessive-compulsive disorder, and the underlying neural mechanism by functional MRI.

DETAILED DESCRIPTION:
All patients underwent a medical evaluation that included physical examination and routine laboratory studies before and after repetitive transcranial magnetic stimulation (rTMS) treatment. Patients were randomly allocated to rTMS group and the sham group. There are about 30 patients in each group. For the first 30 patients, allocation was by coin toss. For the subsequent 30 patients, allocation was according to computer generated random numbers. The decision to enroll a patient was always made prior to randomization. Patients were studied using a double-blind design. Study participants, clinical raters, and all personnel responsible for the clinical care of the patient remained masked to allocated condition and allocation parameters. Only rTMS administrators had access to the randomization list; they had minimal contact with the patients, and no role in assessing the Yale-Brown Obsessive Compulsive Scale(Y-BOCS). Each patient would be treated for continuous 15 days by rTMS.

Before the rTMS treatment, Y-BOCS, Padua Inventory-Washington State University Revision(PI-WSUR), Hamilton Depression Scale(HAMD-17) and Hamilton Anxiety Scale (HAMA-14) were obtained by a trained investigator to assess baseline severity of and other symptoms. The patients had receiving a battery measure of neuropsychological tests (standardized tests to investigate their cognitive problems, anxiety and depressive symptoms in daily life), magnetic resonance imaging scan in multimodalities, electroencephalography (EEG), event-related potentials during stop signal test and task switch paradigm record.

After the last treatment, Y-BOCS, PI-WSUR, HAMD-17 and HAMA-14 were obtained, as well as the Global Index of Safety to assess adverse events of the treatment. Patients were instructed to focus their answers on the past 15 days. The patients had also receiving a battery measure of neuropsychological tests, magnetic resonance imaging scan in multimodalities, and EEG record.

A month after the last treatment, participants were interviewed to obtain the Y-BOCS, PI-WSUR, HAMD-17 and HAMA-14. They were instructed to focus their answers on the past week. Additionally, they were also asked to assess the battery of neuropsychological tests, and have magnetic resonance imaging scan in multimodalities, and EEG record. Afterwards, they were unblinded by the study coordinator.

ELIGIBILITY:
Inclusion Criteria:

Patients met diagnostic criteria for obsessive-compulsive disorder using The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)，confirmed by two clinical psychiatrist.

Y-BOCS total severity scores ≥16（Simple forced obsessions or compulsions ≥ 10），HAMA-14 scores < 14，HAMD-17 scores < 17； Raven's Standard Progressive Matrices（SPM） up to normal levels.

After more than one anti-OCD drugs treatment for 8-10 weeks, no significant improvement in symptoms.

Voluntarily participated and cooperated with the experiment.

Exclusion Criteria:

- History of significant head trauma or neurological disorders. Alcohol or drug abuse. Organic brain defects on T1 or T2 images. History of seizures or unexplained loss of consciousness. Family history of medication refractory epilepsy. recent aggression or other forms of behavioral dyscontrol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Symptom improvement assessed by the Yale-Brown Obsessive Compulsive Scale | up to 1 months
  The Yale-Brown Obsessive Compulsive Scale is a test to rate the severity of obsessive-compulsive disorder symptoms, which measures obsessions separately from compulsions. The scale includes 10 items, the first 5 items are evaluated obsessions, the rest are assessments compulsions. Each item 0-4 points, a total of 40 points. The lower the score, the better the outcome.

SECONDARY OUTCOMES:
Stop-Signal Task | pre-treatment; 1 day post-treatment
  Stop-Signal Task is a typical paradigm for measuring response inhibition and contains three indicators: Stop-signal reaction time (SSRT), the lower the SSRT value, the better the inhibition of reaction; Go task reaction time (GORT), GoRT is usually used in combination with SSRT to reveal the impaired of response inhibition; Stop-signal delays (SSD), SSD value increases, more difficult to inhibit successfully.
Task Switch | pre-treatment; 1 day post-treatment
  Task Switch is a paradigm for measuring cognitive flexibility, which involves the ability to unconsciously shift attention between one task and another and contains two indicators: task repeat and task switch.
Wisconsin CardSorting Test | pre-treatment; 1 day post-treatment
  The Wisconsin Card Sorting Test is a cognitive neuropsychological test, used to determine the abilities of human abstraction, concept formation, working memory and cognitive flexibility. Test measures a total of five indicators: Correct Response, Total Errors, Perseverative Responses, Perseverative Errors and Trials to complete 1st cat.
Hanoi Tower | pre-treatment; 1 day post-treatment
  Hanoi Tower is a test of planning and problem solving, that contains four indicators: total movement, Latency, 1st move reaction time and total reaction time.
Symptom improvement assessed by the Padua Inventory-Washington State University Revision | up to 1 months
  The Padua Inventory-Washington State University Revision is a self-rating scale for the severity of symptoms，that contains 5 subscales, 35 items. Each item 0-4 points, a total of 140 points. The lower the score, the better the outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Medical University, Hefei, Anhui, China